CLINICAL TRIAL: NCT01172249
Title: Non-inferiority Study of the Glucosamine Sulfate + Chondroitin Sulfate Association Capsule in Comparison to the CONDROFLEX® Product in Osteoarthrosis of the Knee
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mantecorp Industria Quimica e Farmaceutica Ltd. (Industry)
Responsible Party: Celso Pereira Sustovich, Medical Director, Mantecorp Industria Quimica e Farmaceutica Ltd.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GLI/P/09-1
Record Dates: First submitted 2010-05-26; First posted 2010-07-29 (Estimated); Last update posted 2010-07-29 (Estimated); Status verified 2010-07

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis; Knee; Glucosamine; Chondroitin
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Glucosamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glucosamine-Chondroitin Mantecorp (Experimental): 1 capsule three times daily before meals (drug test - glucosamine sulfate 500 mg + sodium chondroitin sulfate 400 mg - Mantecorp)
  Interventions: Drug: Glucosamine sulfate + chondroitin sulfate - MANTECORP
- Condroflex (Active Comparator): 1 capsule three times daily before meals (reference medication - glucosamine sulfate 500 mg + sodium chondroitin sulfate 400 mg - Condroflex ®).
  Interventions: Drug: Glucosamine sulfate + chondroitin sulfate - CONDROFLEX

INTERVENTIONS:
Drug: Glucosamine sulfate + chondroitin sulfate - MANTECORP — 1 capsule three times daily before meals (glucosamine sulfate 500 mg + sodium chondroitin sulfate 400 mg).
  Arms: Glucosamine-Chondroitin Mantecorp
Drug: Glucosamine sulfate + chondroitin sulfate - CONDROFLEX — 1 capsule three times daily before meals (glucosamine sulfate 500 mg + sodium chondroitin sulfate 400 mg).
  Other Names: Condroflex ®
  Arms: Condroflex

SUMMARY:
This is an open, prospective, randomized, controlled, parallel, multicenter, non-inferiority study in 250 individuals (125 individuals per group), with 204 evaluable patients with clinical and radiological diagnosis of osteoarthritis of the knee.

Individuals will be randomized to receive during 180 days the test drug(glucosamine sulfate 500 mg + sodium chondroitin sulfate 400 mg - Mantecorp) or the reference medication (glucosamine sulfate 500 mg + sodium chondroitin sulfate 400 mg - Condroflex®).

Efficacy will be evaluated through the clinical picture, pain visual analog scale, swelling, stiffness in the joint, consumption of paracetamol and quality of life.

The safety assessment will be done by monitoring the incidence of adverse events and their relation to the treatment.

DETAILED DESCRIPTION:
This is an open, prospective, randomized, controlled, parallel, multicenter, non-inferiority study in 250 individuals (125 individuals per group), with 204 evaluable patients with clinical and radiological diagnosis of osteoarthritis of the knee.

The subjects in this study are immunocompetent men and women, aged between 55 and 80 years, diagnosed with osteoarthritis of the knee.

The inclusion will be competitive.

Individuals who qualify in the screening period will be randomized to receive during 180 days one of the following regimens below:

* Therapeutic regimen A: one capsule T.I.D. before meals (drug test - glucosamine sulfate 500 mg + sodium chondroitin sulfate 400 mg - Mantecorp)
* Therapeutic regimen B: one capsule T.I.D. before meals (reference medication - glucosamine sulfate 500 mg + sodium chondroitin sulfate 400 mg - Condroflex®).

Efficacy will be evaluated through the clinical picture, pain visual analog scale, swelling, stiffness in the joint, consumption of paracetamol and quality of life.

The safety assessment will be done by monitoring the incidence of adverse events and their relation to the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Individuals must have 55-80 years of age, of both sexes and all races.
* Individuals diagnosed with osteoarthritis in the knee with grades 2 to 3 according to the scale of Kellgren / Lawrence [K / L], in conjunction with the measurement of Joint Space Width (JSW), which considers the joint space width, confirmed by radiological examination (s) of the knee (s) affected (s).

Grade 1: doubtful narrowing of joint space and possible osteophyte edge Grade 2: defined osteophytes, moderate joint space narrowing Grade 3: moderate multiple osteophytes, definite reduction in joint space, some sclerosis and possible deformity of bone contour Grade 4: large osteophytes, marked joint space narrowing, severe sclerosis and definite deformity of bone contour

* Individuals with the capacity to provide a written informed consent, understand and respond to the questionnaires during the study about their disabilities and also with a willingness to adhere to treatment and attend the scheduled appointments for the study.
* Persons who have observed the period of wash-out of the drugs listed in question Prohibited Medication

Exclusion Criteria:

* Individuals with a history of hypersensitivity to glucosamine sulfate and chondroitin sulfate or any of the components of the formula
* Individuals who have used any drug in research within the last 30 days
* Individuals with uric acid greater than or equal to 6 mg/dL for women and 7 mg/dL for men or a previous diagnosis of gout and/or on hypouricemic medication
* Individuals who are in physical therapy
* Individuals with bilateral osteoarthritis, in whom the classification of one of the knees does not fit into grade 2 or 3, according to the scale Kellgren / Lawrence (K/L) together with the measure of Joint Space Width (JSW)
* Individuals being treated with glucocorticoid infiltration, or who have injected hyaluronic acid in the joint
* Individuals who underwent arthroplasty in any location to be evaluated
* Individuals with thyroid dysfunctions that are not controlled (these can only be included in the presence of a normal TSH)
* Subjects with decompensated type 2 diabetes mellitus (diagnosed by examination glycated hemoglobin, which should be below 7.5%)
* Individuals with infection (known or suspected) in the joints that require therapy with systemic antibiotics
* Individuals with significant diseases or clinically significant disorder which, according to the investigator, could interfere with the study or require treatment that might interfere with assessment of efficacy and / or safety
* Individuals who have knowledge of being HIV positive or are immunocompromised
* Patients who need to use some of the medications listed in item Forbidden Medication
* Individuals with other neurological or orthopedic alteration that affects the lower limbs
* Individuals with a BMI (Body Mass Index) greater than 27
* Individuals should not initiate physical activity after the inclusion of the study. If they are already doing regular activities before entering the study, the patient may be included as long as he keeps the activities
* Individuals with kidney disease.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)

PRIMARY OUTCOMES:
WOMAC Index | 180 days
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is a set of standardized questionnaires used by health professionals to evaluate the condition of patients with osteoarthritis of the knee and hip.
Paracetamol use | 180 days
  Another primary outcome measure is the frequency of use of analgesic medication (paracetamol).
Adverse events | 180 days
  Adverse events related to the reference and the test drug will be recorded and used as another primary outcome measure.

SECONDARY OUTCOMES:
Subjective assessment of response to therapy by the investigator and patient | 180 days
  Subjective criteria for evaluating effectiveness:
  Edema - will be evaluated according to the opinion of the physician using the Visual Analogue Scale (VAS).
  Pain - will be assessed according to the opinion of the patient using a visual analog scale (VAS).
  Stiffness in the joint - will be evaluated via the diary and through the patient's opinion also using the Visual Analogue Scale (VAS)
Subjective evaluation of tolerability graded as excellent, good, regular or poor | 180 days
  Subjective evaluation of tolerability to the test and reference drugs will be used as secondary outcome measures. Tolerability will be classified as:
  * Excellent: absence of adverse events;
  * Good: adverse events can be easily tolerated;
  * Regular: adverse events can be tolerated and that do not lead to discontinuation of treatment;
  * Poor: adverse events require treatment discontinuation.